CLINICAL TRIAL: NCT02252913
Title: A Phase Ib, Open-label Study of Safety and Pharmacokinetics of Volitinib in Combination With Docetaxel in Patients With Advanced Gastric Cancer
Brief Title: A Study of Safety and Pharmacokinetics of Volitinib With Docetaxel in Patients With Advanced Gastric Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hutchison Medipharma Limited (Industry)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Organization: Hutchmed (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 2014-504-00CH1
Record Dates: First submitted 2014-09-16; First posted 2014-09-30 (Estimated); Last update posted 2016-04-08 (Estimated); Status verified 2016-04

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — 1-(1-(imidazo(1,2-a)pyridin-6-yl)ethyl)-6-(1-methyl-1H-pyrazol-4-yl)-1H-(1,2,3)triazolo(4,5-b)pyrazine; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Volitinib+docetaxel (Experimental): Dose escalation stage: oral administration, Volitinib 600mg/800 QD + docetaxel 75mg/m2.
  If the dose of docetaxel 75mg/m2 is not tolerable, docetaxel dose will be reduced to 60mg/m2 while keep volitinib at 600mg QD as the initial dose. Volitinib dose escalation will be re-started and end at the dose of 800mg QD.
  Dose expansion Stage:Volitinib with docetaxel. Use the prefer dose from escalation stage
  Interventions: Drug: Volitinib; Drug: Docetaxel

INTERVENTIONS:
Drug: Volitinib — oral administration
  Other Names: HMPL-504
Drug: Docetaxel — intravenous injection
  Other Names: Taxotere

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of volitinib in combination with docetaxel in patients with locally advanced or metastatic gastric cancer and to determine the Maximum tolerated dose (MTD) and/or recommended phase II dose (RP2D) of volitinib in combination with docetaxel.

DETAILED DESCRIPTION:
This is a phase Ib, open-label study.

There are two stages to this study: a dose-escalation stage and a dose-expansion stage. Approximately 40-50 patients will be enrolled in this two-stage study, about 12-18 patients in the dose-escalation stage and approximately 30 patients in the dose-expansion stage.

Dose escalation stage

Gastric cancer patients who failed the first line therapy (no matter the cMet status) who meet the eligibility criteria will be enrolled into this stage.

Cohort 1: Volitinib 600mg QD + docetaxel 75mg/m2 Cohort 2: Volitinib 800mg QD+ docetaxel 75mg/m2 The conventional 3+3 design (3 patients per dose cohort, with the potential to add additional 3 patients to the same cohort to further evaluate toxicity) will be applied for dose escalation and MTD or RP2D determination. Each treatment cycle will be composed of 3 weeks or 21 days. Dose escalation and entry of the next cohort will occur only after acceptable tolerance has been demonstrated throughout the entire Cycle1.

Dose expansion Stage

Additional patients will be enrolled at the MTD or RP2D to further refine the safety, tolerability, PK, and efficacy at this dose. Patients will be limited to the metastatic / locally advanced gastric cancer patients who failed the first therapy and with positive cMet test results. Patients will be divided into two treatment groups according their c-Met test results:

Group A: FISH + , IHC -/+(about 15 patients) Group B: IHC+ and FISH- (about 15 patients)

ELIGIBILITY:
Inclusion Criteria:

1. Signed Informed Consent Form
2. Age ≥18 years
3. Histologically or cytologically documented, locally advanced, or metastatic gastric cancer patients who have failed the first line platinum and fluoropyrimidine based treatment. Adjuvant or neoadjuvant chemotherapy will be considered as first line treatment for advanced disease if disease progression occurred during or within 6 months of treatment.
4. In the dose expansion stage, patients must have positive cMet test results by a central laboratory
5. Absolute neutrophil count (ANC) ≥ 1.5x109/L, hemoglobin ≥ 9 g/dL and platelet count ≥ 100x109/L
6. Total bilirubin ≤ULN; SGOT (AST), SGPT (ALT), ≤ 1.5xULN; alkaline phosphatase (ALP) ≤ 2.5xULN
7. Serum creatinine <1.5xULN or creatinine clearance ≥50mls/minute; confirmation of creatinine clearance is only required when creatinine is >1.5 ULN
8. International normalized ratio (INR) ≤1.5xthe ULN or activated partial thromboplastin time (aPTT) ≤1.5xthe ULN. The INR applies only to patients who do not receive therapeutic anti-coagulation.
9. Evaluable disease at dose escalation stage and measurable disease at dose expansion stage per RECIST v1.1
10. ECOG performance status of 0, or 1
11. Expected survival > 3 months
12. Male or female patients of child-producing potential must agree to double barrier contraception, condoms, intrauterine device (IUD), or contraceptives or other effective avoidance of pregnancy measures during the study and for 90 days after the last dose of treatment
13. Female patients of child-producing potential must have a negative pregnancy test prior to start of dosing or must have evidence of non-childbearing potential by fulfilling one of the following criteria at screening:

    * Post-menopausal defined as aged more than 50 years and amenorrhoeic for at least 12 months following cessation of all exogenous hormonal treatments
    * Documentation of irreversible surgical sterilisation by hysterectomy, bilateral oophorectomy or bilateral salpingectomy but not tubal ligation
    * Women under the age of 50 years would be considered postmenopausal if they have been amenorrhoeic for 12 months or more following cessation of exogenous hormonal treatments and with LH and FSH levels in the post-menopausal range for the institution.
14. Patients with known tumor thrombus or deep vein thrombosis (DVT) are eligible if stable on low molecular weight heparin (LMWH) for ≥4 weeks.

Exclusion Criteria:

1. Prior taxane or cMet inhibitor therapy for advanced disease. Prior taxane containing regimen as adjuvant or neoadjuvant therapy can be allowed provided relapse occurred at least 6 months after therapy
2. Co-existing malignancy or malignancies diagnosed within the last 3 years other than Gastric with the exception of skin basal cell carcinoma or cervical cancer in situ at dose expansion stage.
3. Any anti-cancer therapy, including, but not limited to chemotherapy, hormonal therapy, target therapy, immunotherapy, biologic therapy, radiotherapy, or herbal therapy within 3 weeks prior to initiation of study treatment with the following exceptions:

   * Hormone-replacement therapy or oral contraceptives
   * Palliative radiation to bone metastases 2 weeks prior to Day 1
4. Strong inducers or inhibitors of CYP3A4 or strong inhibitors of CYP1A2 within 2 weeks before the first dose of study treatment (3 weeks for St John's Wort). See appendix 5
5. Adverse events from prior anti-cancer therapy that have not resolved to CTC AE Grade 1, except for alopecia
6. Clinically significant active infection
7. Known clinically significant history of liver disease, including viral or other hepatitis , current alcohol abuse, or cirrhosis
8. Known human immunodeficiency virus（HIV）infection
9. Pregnant or lactating women
10. NYHA Class II or greater congestive heart failure
11. History of myocardial infarction, unstable angina, stroke or transient ischemic attack within 6 months prior to study entry , or cardiac ventricular arrhythmias requiring medication
12. Currently receiving treatment with therapeutic doses of warfarin sodium. Low molecular weight heparin (LMWH) is allowed
13. Brain metastasis or spinal cord compression not definitively treated with surgery and/or radiation, or previously treated CNS metastases or spinal cord compression without evidence of stable disease (clinically stable imaging) for ≥ 14 days. Current leptomeningeal metastases.
14. Inability to take oral medication, prior surgical procedures (except prior total or partial gastrectomy) or serious gastrointestinal disorders such as dysphagia and active peptic ulcer disease that may affect drug absorption in the opinion of the investigator
15. Inability to comply with study and follow-up procedures
16. Known hypersensitivity to taxanes, and/or any components of Volitinib tablet or docetaxel formulation components (eg, polysorbate 80).
17. More than grade 2 peripheral neuropathy or grade 2 peripheral neuropathy with pain.
18. Any other diseases, metabolic dysfunction, physical examination findings, or clinical laboratory finding that, in the investigator's opinion, may give reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that may affect the interpretation of the results or may render the patient at high risk from treatment complications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2014-09; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
safety and tolerability | 21days
  * Incidence and nature of DLTs
  * Incidence and severity of AE/SAEs

SECONDARY OUTCOMES:
PK parameters | 22 days
  * Area Under Curve (AUC)
  * Maximum plasma concentration (Cmax)
  * Clearance (CL/F)
  * Volume of distribution (Vd/F)
  * Other parameters, such as accumulation ratio, elimination half-life

CONTACTS AND LOCATIONS:
Overall Officials: Jin Li, Prof., Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided